CLINICAL TRIAL: NCT00817830
Title: Cardiovascular Safety Evaluation in Patients With Coronary Artery Disease During Physical Effort After Use Lodenafil Carbonate
Brief Title: Cardiovascular Safety Study of Lodenafil Carbonate in Patients With Coronaropathy During Physical Effort
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in patient recruitment
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Dr. Jorge Barros Afiune, Cristália Pordutos Químicos Farmacêuticos Ltda
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CRIST001
Record Dates: First submitted 2008-12-05; First posted 2009-01-07 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2011-06

CONDITIONS: Erectile Dysfunction; Coronaropathy
Keywords: Coronaropathy; lodenafil carbonate; Erectile dysfunction; Treatment; QT interval; Phosphodiesterase inhibitors; Cardiac arrhythmia; Effort testPhosphodiesterase 5 inhibitors; Cardiovascular test
MeSH Terms: conditions — Erectile Dysfunction; Arrhythmias, Cardiac | interventions — lodenafil carbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lodenafil carbonate (Experimental): Evaluate cardiovascular safety of lodenafil carbonate in patients with coronary artery disease undergoing physical effort, before and after using lodenafil carbonate.
  Interventions: Drug: lodenafil carbonate

INTERVENTIONS:
Drug: lodenafil carbonate — Patients will do a cardiopulmonary exercise test after placebo administration. Seven days later, a new cardiopulmonary test should be done using lodenafil carbonate, 80mg, orally.
  Other Names: Helleva

SUMMARY:
The purpose of this study is to assess the safety of lodenafil carbonate in patients with coronaropathy, evaluating the response of the body facing physical effort, including both heart and respiratory components, with and without use of lodenafil carbonate 80mg.

DETAILED DESCRIPTION:
Phosphodiesterase 5 inhibitors (iPDE5) are effective drugs to treat erectile dysfunction (ED).

ED is linked to several factors, like advanced age and diabetes as predominant in its incidence. In addition, ED can be an early manifestation of cardiovascular diseases.

Among the iPDE5 existing in the Brazilian market there is a new molecule which called lodenafil carbonate. It was recently approve and release for use in Brazil, and has similar effectiveness and adverse reactions comparing with other drugs from the same family.

The molecule was evaluated with respect to possible changes in heart rate, blood pressure and QT interval, and the results point out excellent cardiovascular safety profile.

There is a corelated incidence between patients with coronary artery disease and erectile dysfunction. Although patients with stable angina and, under appropriate clinical treatment did not show increase in cardiovascular risks during sexual intercourse, the increased incidence of erectile dysfunction in this population determines a specific group of patients with high potential for use iPDE5.

Therefore it is essential that any new phosphodiesterase 5 inhibitors should be evaluated in patients with coronary artery disease, especially in heart rate, during physical effort.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease with obstruction <70%, confirmed by prior catheterization, stable patient, and have already showed an acute event (unstable angina or myocardial infarction, according to the guidelines of the Brazilian Society of Cardiology) for at least 6 months;
* Age ≥ 18 and ≤ 60;
* Men;
* Stable for 6 months, regardless of previous myocardial infarction or revascularization;
* ejection fraction of doppler echocardiography ≥ 50%.

Exclusion Criteria:

* Use of nitrate;
* Use of bronchodilators;
* Smoking current period or in less than 6 months;
* Hemoglobin <10 g / dL;
* Systolic pressure> 160 mm Hg and <100 mmHg;
* Diastolic pressure> 110 mm Hg and <60 mmHg;
* Body mass index (BMI)> 30;
* Symptomatic peripheral artery disease;
* Event of angina or AMI, at any time, whether I've done some examination or not;
* Finger tip blood glucose < 70 and > 200mg/dL at the time of examination;
* Chest injury > 50%;
* Triple arterial injury with surgery indication;
* Moderate or severe chronic obstructive pulmonary disease (COPD) confirmed by spirometry;
* Pulmonary hypertension with pressure > 35mmHg confirmed by doppler echocardiography;
* Moderate or important aortic and/or mitral valvulopathy confirmed by doppler echocardiography;
* Changes in enzyme markers (Troponin I) after the first test;

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05; Study Completion 2009-10

PRIMARY OUTCOMES:
Evaluate changes in effort test showing the safety of lodenafil carbonate in patients with coronaropathy. | july 2009

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Franken, Doctor, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil